CLINICAL TRIAL: NCT05087732
Title: A Prospective, Triple Blinded, Randomized, Controlled Clinical Study of the Effectiveness and Safety of STYLAGE® M LIDOCAINE Versus STYLAGE® M in Filling Nasolabial Folds
Brief Title: Effectiveness and Safety of STYLAGE® M LIDOCAINE Versus STYLAGE® M in Filling Nasolabial Folds
Acronym: MLIDOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: VIV-STYL-LIDO-01
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Aging
Keywords: hyaluronic acid; Nasolabial Folds; Injection; Healthy subjects; Prospective; Randomized; Pain; Within-subjects
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Within-subject study with treatment of one nasolabial fold with STYLAGE® M and STYLAGE® M Lidocaïne of the other nasolabial fold
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treating investigators (Injectors) , subjects, blinded live evaluator and Independant Photographic reviewer are blinded.
  The product name will not be printed on the labels of investigational device (outside boxes, blisters and syringes )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stylage® M Lidocaïne (Experimental): STYLAGE® M Lidocaine is a hyalorunic acid injectable gel with Lidocaine hydrochloride whose intended purpose is the filling of skin depressions on the face by dermal injection.
  Interventions: Device: STYLAGE® M Lidocaïne; Device: STYLAGE® M
- Stylage® M (Active Comparator): STYLAGE® M Lidocaine is a hyalorunic acid injectable gel whose intended purpose is the filling of skin depressions on the face by dermal injection.
  Interventions: Device: STYLAGE® M Lidocaïne; Device: STYLAGE® M

INTERVENTIONS:
Device: STYLAGE® M Lidocaïne — Up to 2 mL will be injected at Day 0 on a nasolabial fold and, if required, up to 1 mL could be injected 14 days after on the same nasolabial fold (touch-up).
Device: STYLAGE® M — Up to 2 mL will be injected at Day 0 on a nasolabial fold and, if required, up to 1 mL could be injected 14 days after on the same nasolabial fold (touch-up).

SUMMARY:
This clinical investigation is designed to compare the STYLAGE® M Lidocaïne to STYLAGE® M in terms of correction of nasolabial folds severity and pain felt by the subject, and to assess and compare the safety and effectiveness of both products.

Subjects with moderate to severe nasolabial folds will receive both treatments in a split-face design at D0, and a touch-up will be done 14 days after if necessary. The subjects will be followed-up over a 12-month period after initial injection.

DETAILED DESCRIPTION:
The study will be prospective, triple-blinded (Subject, Treating Investigator, and Blinded Live Evaluator),randomized,within-subjects (split-face),active-controlled, monocenter with blinded subjects and evaluators assessing the efficacy , safety and pain of STYLAGE® M Lidocaïne and STYLAGE® M in the treatment of nasolabial folds.

Sixty five healthy subjects between the age of 30 and 65, with symetrical moderate to severe nasolabial folds with grade 3 or 4 on both sides on the Wrinkle Severity Rating Scale (WSRS) for nasolabial folds as assessed in live, who have given their informed consent and met all eligibility criteria, will be enrolled.

STYLAGE® M Lidocaïne will be injected in one nasolabial fold (right or left according to the randomization list). STYLAGE® M will be injected in the contralateral nasolabial fold.

A touch-up is possible if required 14 days after. Subjects will be followed up at 14 days, 3, 6 and 12 months timepoints. All the effectiveness and safety evaluations will be done by a Blinded Live Evaluator (BLE) who will be different from the Treating Investigators.

Variation in severity score of nasolabial folds will be assessed in live by the BLE and retrospectively assessed on photographs (2D) by an Independent Photographic Reviewer using the validated 5-point Wrinkles Severity Rating Scale (WSRS) at each time point The subjects and the independent blinded evaluator will assess the overall aesthetic improvement level of the face, for each side independently, at each time point after treatment initiation The subjects will be asked to score the pain felt during injection, and 5, 15 and 30 minutes after injection on a Visual Analog Scale .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject.
2. Age: between 30 and 65 years.
3. Subject with right and left NLF rating grade 3 or 4 (Moderate or Severe) on the Wrinkle Severity Rating Scale (WSRS), as assessed by a Blinded Live Evaluator.
4. Subject having the same WSRS grade on both NLFs (i.e., symmetrical NLFs).
5. Subject with marionette's lines that do not require to be treated in addition to nasolabial folds, according to the Blinded Live Evaluator.
6. Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures (i.e., dermal fillers, toxin treatments, facial ablative or fractional laser, microdermal abrasion, chemical peels, non-invasive skin-tightening) below the level of the lower orbital rim, for the duration of the study.
7. Subjects agreeing not to take Anti-histamines within 2 weeks prior to touch-up visit
8. Subject able to comply with protocol requirements and to complete all required visits.
9. Subject, psychologically able to understand the study related information and to give a written informed consent.
10. Subject having given freely and expressly his/her informed consent to participate in the study, and use of data privacy, prior to any study-related procedure being performed.
11. Subject agreeing to have photographs taken.
12. Female of childbearing potential must have a negative urinary pregnancy test (UPT) at Visit 1 and practice a reliable method of contraception throughout the study, and for at least 12 weeks prior to study enrolment.
13. Subject affiliated to a health social security.

Exclusion Criteria:

1. Subject presenting any symptom which can be related to a medical condition that is likely to make the subject not being compliant with the study schedule, at the discretion of the investigator
2. Pregnant or breastfeeding woman or planning a pregnancy during the study.
3. Had prior surgery in the mid- and/or lower-face area, including the nasolabial fold(s), or has a permanent implant or graft in the mid- and/or lower-face area, or a tattoo, a scar, moles, or anything that could interfere with effectiveness assessments. (NOTE: Rhinoplasty is permitted if the procedure was ≥ 12 months prior to study enrolment).
4. Subject in a social or sanitary establishment.
5. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
6. Subject participating to another research on human beings or who is in an exclusion period of one.
7. Subject having received 4500 euros indemnities for participation in researches involving human beings in France in the 12 previous months, including participation in the present study.
8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
10. Subject with a past history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats with cardiac localisation.
11. Subjects suffering from porphyria.
12. Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…). Subject with recurrent herpes is not eligible even if asymptomatic at time of inclusion.
13. Subject having history of severe allergy or anaphylactic shock including hypersensitivity to hyaluronic acid, to gram positive bacterial proteins, to lidocaine or antiseptic solution or amide type local anaesthetics.
14. Subject predisposed to develop keloids or hypertrophic scarring.
15. Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
16. Subject having received treatment with a laser, a dermabrasion, a surgery, a peeling or other ablative procedure below the inferior orbital rim within the past 6 months prior to study start.
17. Subject having received injection with a resorbable filling product (eg, hyaluronic acid, collagen) below the inferior orbital rim within the past 12 months prior to study start.
18. Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), etc.) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, etc.).
19. Subject having received at any time a treatment with tensor threads below the inferior orbital rim.
20. Subject who received oral surgery (tooth extraction, orthodontia or implantation) within 6 weeks prior to study start or who plans to undergo any of these procedures during the study.
21. Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to study start or planning to change it during the study.
22. Subject using medication such as aspirin, nonsteroidal anti-inflammatory drugs (NSAID) (ibuprofen, naproxen, etc.), antiplatelet agents, anticoagulants, vitamin C or other substances known to increase coagulation time within one week prior to treatment dates.
23. Subject using medication that reduce or inhibit hepatic metabolism (cimetidine, beta-blockers, etc.).
24. Subject undergoing a topical treatment on the test area or a systemic treatment:

    * Anti-histamines during the 2 weeks prior to study start;
    * Immunosuppressors and/or corticoids during the 4 weeks prior to study start;
    * Retinoids during the 6 months prior to study start.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Difference of aesthetic improvement on the Wrinkle Severity Rating Scale (WSRS), | 6 months
  First co-primary endpoint will be the difference of aesthetic improvement on the Wrinkle Severity Rating Scale (WSRS), as evaluated by the BLE, at the side of the face treated with Stylage® M lidocaïne compared to the side of the face treated with Stylage® M, in a double non-inferiority statistical model.
Within-subject difference in injection site pain | immediatly after injection of each side
  Second co-primary endpoint will be the (STYLAGE® M Side - STYLAGE® M lidocaine Side), self-assessed by the subjects on a 100 mm Visual Analogue Scale (VAS), in a superiority statistical model.

SECONDARY OUTCOMES:
WSRS change from baseline | 4 days, 3, and 12 months after baseline
  WSRS change from baseline as assessed by the Blinded Live Evaluator (BLE)
WSRS change from baseline on photographs | 14 days, 3, 6, and 12 months after baseline
  WSRS change from baseline as assessed by an Independent Photographic Reviewer (IPR), on photographs.
Responder rate for WSRS in live | 14 days, 3, 6, and 12 months after baseline
  Responder rate for WSRS , as assessed by the BLE. A responder is defined as a subject with at least 1-point improvement from baseline on the WSRS.
Responder rate for WSRS on photograph | 14 days, 3, 6 and 12 months after baseline
  Responder rate for WSRS , as assessed by an Independent Photographic Reviewer (IPR), on photographs.
Global Aesthetic Improvement assessed by the BLE | 14 days, 3, 6, and 12 months after baseline
  Global Aesthetic Improvement assessed by the BLE on the Global Aesthetic Improvement Scale (GAIS).
Global Aesthetic Improvement assessed by the Subject | 14 days, 3, 6, and 12 months after baseline
  Global Aesthetic Improvement assessed by the Subject on the Global Aesthetic Improvement Scale (GAIS).
Proportions of GAIS responders assessed by the BLE | 14 days, 3, 6, and 12 months after baseline.
  Proportions of GAIS responders defined as subjects with a GAIS score " Improved ", " Much Improved ", or " Very Much Improved ", as assessed by the BLE
Proportions of GAIS responders assessed by the subjects | 14 days, 3, 6, and 12 months after baseline.
  Proportions of GAIS responders defined as subjects with a Global Aesthetic " Improved ", " Much Improved ", or " Very Much Improved ", as assessed by the subjects
Subject Satisfaction questionnaire | 14 days, 3, 6, and 12 months
  Proportion of subjects either " Somehow satisfied ", " Satisfied ", or " Very Satisfied ", as assessed by the subjects
Injection Site Pain self-assessed by the subjects (touch-up) | immediatly after touch-up injection
  Injection Site Pain during injection self-assessed by the subjects of each side during optional touch-up treatment (VAS 100mm).
Injection Site Pain self-assessed by the subjects (initial and touch-up) | 5, 15, and 30 minutes post-injection
  Injection Site Pain self-assessed by the subjects at during initial and optional touch-up treatment.
Proportion of subjects who reported at least 10 mm, 20 mm, and 30 mm less VAS pain (initial and touch-up). | immediately after injection, and at 5, 15, and 30 minutes after each injection
  Proportion of subjects who reported at least 10 mm, 20 mm, and 30 mm less VAS pain associated with injections of Stylage® M Lidocaïne compared to Stylage® M, immediately after injection (initial and touch-up).
Proportion of subjects that reported at least half less VAS pain (initial and touch-up) | Immediately after injection, and at 5, 15, and 30 minutes after each injection
  Proportion of subjects that reported at least half less VAS pain associated with injections of Stylage® M Lidocaïne compared to Stylage® M (initial and touch-up).
Injection site reaction and adverse events reporting | up to 12 months
  Product tolerance will be assessed by collection of Injection Site Reactions (ISRs) after each injection session, and Adverse Events throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Siham RHARBAOUI, Principal Investigator — Dermscan Pharmascan
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No